CLINICAL TRIAL: NCT03409419
Title: PET Imaging of the Immune System Using New Nucleotide Analog Probes
Brief Title: PET Imaging of the Immune System Using Analog Probes
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Tesaro, Inc. (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-001172; NCI-2018-01547 (Registry Identifier: CTRP)
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Malignant Melanoma
Keywords: Advanced; Recurrent; Immune Therapy
MeSH Terms: conditions — Melanoma; Recurrence | interventions — Product Labeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre cohort: Each subject will undergo a maximum of two 18F-Clofarabine PET/CT scans with each visit taking up to 4 hours. The 18F-Clofarabine PET/CT scans will be performed before the treatment interventions.
  Interventions: Drug: [18F] CFA
- post cohort: Each subject will undergo a maximum of two 18F-Clofarabine PET/CT scans with each visit taking up to 4 hours. The 18F-Clofarabine PET/CT scans will be performed after the treatment interventions.
  Interventions: Drug: [18F] CFA

INTERVENTIONS:
Drug: [18F] CFA — pilot study to evaluate the bio-distribution of [18F] CFA, a new tracer for imaging the purine nucleoside biosynthetic pathway, before and after immunotherapy treatment in patients with metastatic or recurrent advanced melanoma.
  Other Names: tracer for imaging the purine nucleoside biosynthetic pathway

SUMMARY:
The goal of this proposal is to assess the biodistribution of 18F-Clofarabine, a new tracer developed for use in PET/CT scans. The investigator's hypothesis is this tracer will allow for imaging immune activation in patients with melanoma before and after treatment with immunotherapy.

A maximum of 10 subjects are intended to be included in this study. Each subject will undergo a maximum of two 18F-Clofarabine PET/CT scans, with each visit taking up to 4 hours. The first visit will be prior to the first cycle of immunotherapy treatment, and the second scan will take place 2-4 weeks after the immunotherapy treatment has started.

Prior to the PET scan an IV line will be placed. Blood pressure, heart rate, blood oxygen and ECG will be obtained. Then the 18F-Clofarabine will be injected and the PET/CT scan acquisition started. After a maximum of 120 min of scanning, subjects will undergo again blood pressure, heart rate, blood oxygen and ECG.

DETAILED DESCRIPTION:
This is a non-interventional pilot study dedicated to PET imaging for patients with metastatic or recurrent advanced cancer melanoma before and after immune therapy interventions with an anti-TIM-3 monoclonal antibody, with or without an anti-PD1 antibody.

PET/CT will be used to investigate the bio-distribution of 18F-Clofarabine in patients with advanced or metastatic melanoma before and 2 to 4 weeks after immune system activating interventions, namely an anti-TIM-3 monoclonal antibody, alone or in combination with an anti-PD1 antibody. Clofarabine is a FDA-approved drug for treatment of relapsed or refractory pediatric acute lymphoblastic leukemia (December 2004) and is gaining importance for treating adult patients with acute myeloid leukemia. Despite extensive preclinical toxicity studies and multiple human phase I studies, the exact bio-distribution of Clofarabine remains unknown. The labeling of Clofarabine with 18F allows the in vivo imaging of its bio-distribution using only minimal concentrations of the therapeutically active doses. The radioactive labeling of clofarabine does not change the parent molecule since a 19F present in the parent compound is simply replaced by an 18F.

The investigators hypothesize that imaging the bio-distribution of clofarabine non-invasively will provide insights into the bio-distribution of the drug in vivo. Imaging the bio-distribution of radiolabeled Clofarabine may help to better understand the side effects caused by therapeutic doses. Importantly, the investigators want to understand if interventions activating the immune system impact the bio-distribution of 18F-Clofarabine. This is because the enzyme dCK that is required to activate the prodrug clofarabine is highly expressed in activated immune cells (3).

Dynamic PET/CT imaging with 18F-Clofarabine will be performed in 10 patients with advanced or metastatic melanoma who have progressed following treatment with an anti-PD-1 antibody. 18F-Clofarabine PET/CT scans will be collected before and 2-4 weeks after treatment with an anti-TIM-3 monoclonal antibody, with or without an anti-PD1 antibody. Imaging can be completed without exposing human subjects to any significant risk. It should be noted, that only trace amounts (nano-molar concentrations in saline solution) of the labeled 18F-Clofarabine will be administered intravenously. Thus, mass effects of the drug and any toxic effects can be ruled out. Tracer concentrations in all organs can be quantified non-invasively in organs which may provide insights into the whole-body drug distribution. Investigators have now seen in humans and non-human primates the exact bio-distribution that one would expect with uptake in bone marrow, spleen, LN and, if patients are young, in thymus. Liver uptake is non-specific and likely due to hepatic clearance via biliary system. There is no retention in other organs which does not mean that there is no low background activity. Tracer uptake is proportional to dCK activity in tissues.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria also apply:

1. Subject must be able to tolerate PET/CT (i.e. not claustrophobic and able to remain supine)
2. Subject must be 18 years or older
3. Participation in a main study of anti-TIM-3

Exclusion Criteria:

* Patients who meet the exclusion criteria are excluded from this study. 1. Pregnancy

  1. Women of childbearing potential will have to undergo a pregnancy test that will be provided free of charge.
  2. Current knowledge indicates no confirmed detrimental effects to a developing fetus of radiation doses below 10,000 mrem. The radiation dose received from the study procedure is very small in comparison, however, the exclusion criteria is in place to minimize any potential for exposure of a fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients with advanced or metastatic melanoma who have progressed following treatment with an anti-PD-1 or anti-PD-L1 antibody, who are enrolled in a clinical trial and scheduled to receive an anti-TIM-3 monoclonal antibody, alone or in combination with an anti-PD1 antibody, will be eligible for this study.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
biodistribution of tracer | 6 weeks
  The biodistribution of 18F-Clofarabine in melanoma patients

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, M.D., Principal Investigator — UCLA/Jonsson Comprehensive Cancer Center
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States